CLINICAL TRIAL: NCT05779566
Title: Exploratory Evaluation of the Functional/Emotional Life Characteristics During the First Year of Ongoing Endocrine Adjuvant Treatment With Aromatase Inhibitors in Breast Cancer Patients With Reduced Bone Mineral Density
Brief Title: Evaluation of the Functional/Emotional Life Characteristics of Ongoing EAT in BC Patients With Reduced BMD
Acronym: REBECCA-OST
Status: Completed | Type: Observational
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/005-OST
Record Dates: First submitted 2022-10-07; First posted 2023-03-22 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer; Osteopenia
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases, Metabolic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- OST: Patients with osteoporosis or severe osteopenia defined as having a significantly reduced BMD (T-score equal or lower than -1.5)
  Interventions: Diagnostic Test: bone densitometry
- Mild OST: Patients with mild-to-no reduction of BMD at the same post-treatment time point (T-score higher than -1.5)
  Interventions: Diagnostic Test: bone densitometry

INTERVENTIONS:
Diagnostic Test: bone densitometry — bone densitometry every 6 month

SUMMARY:
Exploratory evaluation of the Functional/Emotional Life characteristics during the first year of ongoing endocrine adjuvant treatment with Aromatase Inhibitors in Breast Cancer patients (BCP) with reduced Bone Mineral Density (BMD)

DETAILED DESCRIPTION:
Many breast cancer therapies cause decreases in bone mineral density (BMD), as a result of oestrogen deprivation, a well-established risk factor for osteopenia (OST), osteoporosis and bone fractures. That leads to breast cancer patients having reduced bone mass, leading to higher risk for bone osteoporosis-related fractures, compared with age-matched healthy women, necessitating routine bone health assessments after a diagnosis of breast cancer. Such treatments include adjuvant endocrine therapies (e.g., tamoxifen and aromatase inhibitors) commonly used for hormone receptor-positive breast cancers, the most common type of breast cancer.

Additionally, chemotherapy or ablation of ovarian function (either medically or surgically) can lead to premature menopause among younger women and further reduce BMD5. Despite the advances in the pharmacology managing cancer treatment-induced osteopenia, the long-term efficacy of drug effects is debatable6 and there are numerous concerns about rare (but significant) side-effects of anti-resorptive drugs, particularly bisphosphonates. Those challenges necessitate additional research for the optimal OST management as a chronic breast cancer comorbidity.

Thus, the elucidation of the precise onset and progress of OST in patients and its interaction with lifestyle and high risk behaviours are now receiving increased research attention, aiming at the identification of novel patient management strategies to alleviate the chronic effects of the condition.

In order to counter the important life-effects of OST in breast cancer patients, current disease management schemes propose the integration of non-pharmacologic measures to maintain (or improve) optimal bone health, such as weight-bearing exercises and calcium and vitamin D supplementation. However, the lack of objective RWD on the effects of increased BMD on lifestyle is a serious challenge for the design of pragmatic and individualized patient management strategies. Indeed, lifestyle advice for increased physical activity are usually generic, lacking disease-specific knowledge, probably affecting the efficacy of exercise interventions. Overall, further evidence is required to optimise antiresorptive treatments, the use and choice of pharmacological agents, the duration of treatment and the potential of interaction with ongoing endocrine treatment.

Thus, the study will conduct the longitudinal comparison of Functional and Emotional Life Indices in Breast Cancer patients exhibiting significant reduction of BMD up to 12 months of adjuvant treatment with aromatase inhibitors, compared against matched BCPs with mild reduction of BMD. The study will use RWD to assess the safety and the effectiveness of aromatase inhibitor adjuvant endocrine therapy, with regards to osteopenia symptomatology over time. The study will consider data from 3 routine clinical evaluations (study month 0, 6 and 12) for the objective evaluation of BMD loss, complemented with continuous REBECCA use for 12 months. The collected data will include:

* Patient-reported measures: Medical and treatment history interview, project-related measurements, health-related quality of life, adjuvant treatment compliance estimation
* Medical examination: Gynecological physical and anthropometric examination, blood sampling, densitometry

For the REBECCA use, the participants will be trained in the use of the monitoring modules of the REBECCA platforms, facilitating the collection of real-world data (12 months). They will return (after 6 months) for a routine medical evaluation of osteopenia-related symptomatology and adjuvant treatment evaluation. They will complete a QoL questionnaire, and perform a structured interview, concerning mainly the appearance of new symptoms and adverse events or signs regarding bone issues, as well as a gynecological exam.

Blood tests will be collected, compliance to treatment will be evaluated and treatment satisfaction will be assessed.

The meeting will be repeated at 12 months, including a BMD examination

ELIGIBILITY:
Inclusion Criteria:

* Before patient registration, written informed consent must be given according to national and local regulations.
* Participants have had histologically proven stage I-III breast cancer undergoing endocrine treatment (with or without prior chemotherapy) no more than 12 months prior to randomization.
* Be between 18 and 75 years of age.
* Have increased life expectancy beyond the initial 3 months post-treatment initiation.
* Have the ability to understand protocol, participate in testing and willingness to sign a written informed consent.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Exclusion Criteria:

* Patients already diagnosed with Osteopenia/Osteoporosis and already receiving BMD treatment (bisphosphonates or denosumab)
* Patients already diagnosed with osteopenia/osteoporosis who have already suffered a bone event related to decreased BMD
* Patients that are not willing to sign an informed consent form

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study participant recruitment pool will be the whole population of BCPs undergoing endocrine adjuvant treatment (aromatase inhibitors) in the Oncology Department at Hospital Clínico de Valencia (Spain). As part of the ongoing patient follow-up, potential candidates with significant or milder reductions in BMD will be identified at study inclusion (early stages of adjuvant treatment period) based on comparisons with standard population BM measures (i.e., densitometry examination outcome: T-score lower than -1.0211). At this point, appropriate patients interested in the study will be informed about the study and written consents will be obtained.
  All the potential participants will be female due to the nature of Breast Cancer
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Bone mineral density (BMD) | 1 year
  Chronic osteopenia, as a result of significant reduction of BMD, is expected to significantly negatively affect Functional Life characteristics in BCPs undergoing adjuvant endocrine aromatase inhibitors treatments in comparison to those with milder symptomatology.
  The association of the long-term outcomes of the PROM Index with the trajectory of reduced BMD-related symptomatology, as well as the Functional Life Index progression will be examined as an estimate of the safety and the effectiveness of the aromatase inhibitor adjuvant endocrine therapy.
  It is expected that the severity of reduced BMD-related symptomatology is associated with further deterioration of the Functional Life Index.
  Units: gr/cm^2

SECONDARY OUTCOMES:
Adjuvant treatment compliance | 1 year
  Adjuvant treatment compliance estimation (scale scored from 1 to 10)
Weight | 1 year
  Weight measurement (kg) as part of the anthropometric examination
Height | 1 year
  Height measurement (cm) as part of the anthropometric examination
C-Telopeptide concentration | 1 year
  C-Telopeptide concentration (pg/mL) from the blood samples extracted over the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://rebeccaproject.eu/

DOCUMENTS (1):
  • Informed Consent Form (2022-01-05): https://cdn.clinicaltrials.gov/large-docs/66/NCT05779566/ICF_000.pdf